CLINICAL TRIAL: NCT01100879
Title: Randomised Controlled Open-label Study to Evaluate Efficacy & Safety of Intravenous Ferric Carboxymaltose Versus no Treatment in Anaemic Subjects With Multiple Myeloma & Iron Restricted Erythropoiesis Receiving Chemotherapy
Brief Title: Ferric Carboxymaltose for Treatment of Anaemia of Cancer in Subjects With Multiple Myeloma Receiving Chemotherapy
Acronym: AOC-MM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of Recruitment
Sponsor: Vifor Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FER-AOC-MM
Record Dates: First submitted 2010-03-29; First posted 2010-04-09 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2011-06

CONDITIONS: Iron-Deficiency Anemia
Keywords: Anemia; Lymphoproliferative Disorders; Chemotherapy; ferric carboxymaltose; iron
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia; Lymphoproliferative Disorders | interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferric carboxymaltose (Active Comparator): Subjects will receive a total dose of 1,000 mg iron as FCM on the day of the next scheduled chemotherapy cycle after randomisation or continuous chemotherapy. In subjects with weight ≤66 kg, the first dose iron will be 500 mg; the second dose (500 mg) will be administered on the visit 3 (week 2).
  Interventions: Drug: Ferric carboxymaltose
- Local standard of care. (No Intervention): Subjects will be treated according to the local institutional practice.

INTERVENTIONS:
Drug: Ferric carboxymaltose — Subjects will receive a single dose of 1,000 mg iron as FCM infusion at baseline.
  Subjects of bw ≤66 kg will receive a single dose of 500 mg iron as FCM infusion at baseline (Week 0) and at Visit 3 (Week 2).
  Ferric carboxymaltose will be administered on the same day with chemotherapy treatment or within 24 hours before or after the chemotherapy. For subjects with bw ≤66 kg, if no chemotherapy planned for the visit 4 (Week 2), the second FCM dose should be infused independent of chemotherapy.
  Other Names: Ferinject
  Arms: Ferric carboxymaltose

SUMMARY:
Multicentre, randomised, controlled, 2-arm open-label prospective pilot study to evaluate efficacy and safety of ferric carboxymaltose (FCM) in treatment of anaemia in subjects with multiple myeloma (MM) initiating chemotherapy. The subjects will be screened for eligibility within 4 weeks prior to inclusion and randomised to receive intravenous infusions of FCM or standard care (the subjects may be treated according to the local institutional practice if requiring symptomatic management of anaemia). Thereafter the visits are scheduled at Weeks 0, 2, 4, 6 and 8.

DETAILED DESCRIPTION:
Patients will be randomised into two groups. One will receive active FCM treatment and the other group will receive local standard of care.

Active treatment group: Subjects will receive a total dose of 1,000 mg iron as FCM on the day of the first scheduled chemotherapy cycle or within 24 hours before or after receiving chemotherapy. In subjects of weight ≤66 kg, the first dose (500 mg) will be administered on the day of the first scheduled chemotherapy cycle and the second dose (500 mg) on the next study visit.

Standard of care group: Subjects will be treated according to the local institutional practice if requiring management of symptomatic anaemia. Intravenous iron should only be used to treat absolute iron deficiency (as defined as ferritin less than the lower limit of normal based on the test reference ranges). Patients with absolute iron deficiency are not eligible for inclusion to the study.

Rescue medication to manage anaemia is permitted in both arms at the discretion of the treating physician and/or per institutional practice.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (male or female) aged ≥18, suffering from a newly diagnosed or progressed/relapsed MM and scheduled to receive anti-myeloma treatment. Progression is defined according to "Uniform Response Criteria for Multiple Myeloma"
* Subjects with progressed/relapsed MM should have had stable disease (during the last 6 months since prior treatment).
* Life expectancy at least 6 months.
* 8.5 g/dL ≤Hb ≤11 g/dL at time of randomisation.
* Iron-restricted erythropoiesis as defined:

  * Stainable iron in bone marrow (BM) combined with transferrin saturation (TSAT) ≤20%, or
  * where the evaluation of stainable iron in BM is not possible or available:
* ferritin >30 ng/mL (women) or >40 ng/mL (men), and
* TSAT ≤20%
* Females of child-bearing potential must have a negative urine pregnancy test at screening.
* Before any study-specific procedure, the appropriate written informed consent must be obtained.

Exclusion Criteria:

* Any anaemia treatment within 4 weeks prior to randomisation (including red blood cell transfusions, treatment with ESA or any oral/parenteral iron preparations).
* Anthracycline containing chemotherapy regimens.
* Subjects weighing <35 kg.
* Folate deficiency (serum-folate <4.5 nmol/L) and/or Vitamin B12 deficiency (serum-cobalamin <145 pmol/L).
* Ongoing haemolysis defined as serum-haptoglobin <0.2 g/L.
* Known chronic renal failure, glomerular filtration rate <30 mL/min/m2.
* Recent (within last 4 weeks) significant bleeding/surgery, defined as drop in Hb of ≥2 g/dL.
* Clinically relevant active inflammatory disease other than MM (according to the judgement of the Investigator).
* Clinically relevant ongoing infectious disease including known human immunodeficiency virus.
* Serum ferritin >600 ng/mL.
* Ongoing significant neurological or psychiatric disorders including psychotic disorders or dementia.
* Significant cardiovascular disease prior to study inclusion including myocardial infarction within 12 months prior to study inclusion, congestive heart failure New York Heart Association Grade III or IV, or poorly controlled hypertension according to the judgment of the Investigator.
* Elevation of liver enzymes (aspartate aminotransferase, alanine aminotransferase) over 3 times above the normal range or known acute hepatic disorder.
* Subject currently is enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study(ies), or subject is receiving other investigational agent(s).
* Subject of child-bearing potential is evidently pregnant (e.g., positive human chorionic gonadotropin test) or is breast feeding.
* Subject is not using adequate contraceptive precautions. Adequate contraceptive precautions are defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intra-uterine devices, sexual abstinence or vasectomised partner. Non-childbearing potential includes being surgically sterilised at least 6 months prior to the study or post-menopausal, defined as amenorrhea for at least 12 months.
* Subject has known sensitivity to any of the products to be administered during dosing.
* Subject will not be available for follow-up assessment.
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in haemoglobin (Hb) from baseline to Weeks 4, 6 and 8 | week 4, 6 and 8 post baseline
  Mean change in Hb from baseline to Weeks 4, 6 and 8 (end of treatment) in the absence of any red cell transfusion or erythropoiesis stimulating agents (ESA) treatment.

SECONDARY OUTCOMES:
Percentage of subjects with blood Hb response of at least 1 g/dL | 12 weeks post baseline
  Percentage of subjects with blood Hb response of at least 1 g/dL in the absence of any red cell transfusion or ESA treatment.
Percentage of subjects with a blood Hb correction to at least 12 g/dL | 12 weeks post baseline
  Percentage of subjects with a blood Hb correction to at least 12 g/dL in the absence of any red cell transfusion or ESA treatment
Time to Hb response defined as increase in Hb equal to or more than 1 g/dL | Baseline until end of study (week 8)
  Median time to Hb response defined as increase in Hb equal to or more than 1 g/dL in the absence of any red cell transfusion or ESA treatment
Subjects receiving red blood cell transfusions or subjects treated with ESA | Baseline until end of study (week 8)
  Proportion of subjects receiving red blood cell transfusions or subjects treated with ESA during the study period
Adverse events | Baseline until end of study (week 8)
  Adverse events: type, nature, incidence and outcome
Transfusion/treatment with ESA | Baseline until end of study (week 8)
  Time to transfusion/treatment with ESA
Change in serum ferritin from baseline to Weeks 2, 4, 6 and 8 | week 2, 4, 6, and 8 post baseline
  Mean change in serum ferritin from baseline to Weeks 2, 4, 6 and 8
Change in transferrin saturation (TSAT) from baseline to Weeks 2, 4, 6 and 8 | week 2, 4, 6, and 8 post baseline
  Mean change in TSAT from baseline to Weeks 2, 4, 6 and 8
Change in serum iron from baseline to Weeks 2, 4, 6 and 8 | week 2, 4, 6, and 8 post baseline
  Mean change in serum iron from baseline to Weeks 2, 4, 6 and 8
Change in endogenous erythropoietin from baseline to Weeks 2, 4, 6 and 8 | week 2, 4, 6, and 8 post baseline
  Mean change in endogenous erythropoietin from baseline to Weeks 2, 4, 6 and 8
Change in blood reticulocyte haemoglobin content/red blood cell size factor from baseline to Weeks 2, 4, 6 and 8 | week 2, 4, 6, and 8 post baseline
  Mean change in blood reticulocyte haemoglobin content/red blood cell size factor from baseline to Weeks 2, 4, 6 and 8
Change in percentage of hypochromic red cells/percentage of low Hb density from baseline to Weeks 2, 4, 6 and 8 | week 2, 4, 6, and 8 post baseline
  Mean change in percentage of hypochromic red cells/percentage of low Hb density from baseline to Weeks 2, 4, 6 and 8
Change in hepcidin from baseline to Weeks 2, 4, 6 and 8 | week 2, 4, 6, and 8 post baseline
  Mean change in hepcidin from baseline to Weeks 2, 4, 6 and 8
Change in interleukin-6 from baseline to Weeks 2, 4, 6 and 8 | week 2, 4, 6, and 8 post baseline
  Mean change in interleukin-6 from baseline to Weeks 2, 4, 6 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Katodritou Eirini, MD, Principal Investigator — Theagenion Hospital, Thessaloniki, Greece; Timothy R Cushway, Study Director — Vifor Pharma, CH-8152 Glattbrugg, Switzerland
Locations (2):
- Hopital Sud, Rennes, France
- Theagenion Cancer Center, Thessaloniki, Greece